CLINICAL TRIAL: NCT05246683
Title: LATIN SHOCK: Registro Latinoamericano de Shock Cardiogénico en el Contexto de Los Sindromes Coronarios Agudos
Brief Title: LATIN SHOCK: Latin American Registry of Cardiogenic Shock in the Context of Acute Coronary Syndrome
Acronym: LATIN-SHOCK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sociedad Argentina de Cardiología (Other)
Responsible Party: Sponsor
Other Study IDs: LATIN SHOCK
Record Dates: First submitted 2021-12-26; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Cardiogenic Shock; Acute Coronary Syndrome
MeSH Terms: conditions — Shock, Cardiogenic; Acute Coronary Syndrome | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cohort: Observational evaluation during the hospital stage on diagnosis, treatment and evolution of patients with cardiogenic shock.
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — registry

SUMMARY:
This is a Registry of the characteristics and clinical evolution of patients admitted for acute coronary syndromes (with or without st segment elevation) who present with cardiogenic shock or develop it during the hospitalization period.

Cardiogenic shock is a rare pathology, but it constitutes the leading cause of mortality in patients hospitalized for acute infarction myocardium. Its incidence ranges between 7 and 10% of the cases of infarction1 and is associated with a mortality of 40-50% despite revascularization and the use of Intra-Aortic Counterpulsation Balloon. Most of the bibliography on this subject is North American and has a lot of years and the one currently published shows mostly the results of different ventricular supports that are not used routinely in our countries. So far there is no record that reports the reality of Latin America. Only in Argentina, a registry has been carried out (Re Na Shock) but more than 5 years have passed since its publication. In the last years have even changed the management guidelines for this pathology and have been published works that could have changed previous behaviors

. This is a project of the Argentine Society of Cardiology to collect data epidemiological and current management of cardiogenic shock in Latin America.

DETAILED DESCRIPTION:
It is an international, multicenter, observational registry of prospective and consecutive patients with cardiogenic shock in the context of acute coronary syndromes, which will last 12 months from its start on December 4, 2021. Coronary Units will be invited to participate from different Latin American countries through the different cardiology societies. It will be assigned to each country and each participant center a number and patients will be entered into the registry in correlative order by center (1-2-3-etc) to maintain the confidentiality of the patients data. Since the patient data will be extracted from the medical records, the records will be anonymous and there will be no follow-up, no informed consent is required. The names of the participating centers of the different countries will appear in a list at the end of the publications, under the collective name of "LATIN Shock group".

Definition of cardiogenic shock (classic): presence of systolic blood pressure

≤ 90 mm Hg for 30 minutes or requirement of vasopressors, inotropics and / or ventricular supports to maintain a blood pressure ≥ 90 mm Hg, associated with signs of hypoperfusion and pulmonary congestion, in the absence of hypovolemia or arrhythmias that justify the clinical picture. A new definition of cardiogenic shock has recently been proposed (SCAI), which includes 5 categories. In this work, patients with cardiogenic shock only those with C, D and E letter will be included.

ELIGIBILITY:
Inclusion Criteria:Patients of both sexes and older than 18 years, admitted to the unit coronary or polyvalent critical care, for an acute coronary syndrome with or without ST-segment elevation presenting cardiogenic shock from the admission or develop it during the hospitalization and that can be followed in its evolution until hospital discharge. -

Exclusion Criteria:Non-ischemic cardiogenic shock (chronic heart failure, myocarditis, sepsis, tachycardiomyopathies, Takotsubo, etc.). Cardiogenic shock A and B of the new SCAI classification

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute cardiac syndrome with or without st elevation and cardiogenic shock as a complication. Includes cardiogenic shock at presentation or during hospitalario period
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-12-18 (Estimated); Study Completion 2022-12-18 (Estimated)

PRIMARY OUTCOMES:
Register through the survey modality the incidence of the clinical characteristics of the patients admitted to the coronary unit with acute coronary syndromes and cardiogenic shock, either from admission or during its in-hospital evolution. | 1 year
  characteristics
To analyze the treatment and diagnostics methods of patients with cardiogenic shock during hospital stay. | 1 year
  treatment
Observe in-hospital clinical evolution and incidence of complications of patients with cardiogenic shock. | 1 year
  evolution

SECONDARY OUTCOMES:
Find predictors of in-hospital mortality. | 1 year
  predictors
To compare the clinical, management and evolution characteristics in the different participating Latin American countries. | 1 year
  compare

CONTACTS AND LOCATIONS:
Overall Officials: Victor M Mauro, md, Study Director — Sociedad Argentina de Cardiologia
Locations (1):
- Sociedad Argentina de Cardiologia, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/83/NCT05246683/Prot_SAP_000.pdf